CLINICAL TRIAL: NCT05548621
Title: A Prospective Study to Evaluate the Implementation of Shared Decision Making Strategy for Renal Cell Cancer (RCC)
Acronym: SDM-RCC
Status: Recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Cato Bresser, Coordinating Investigator, St. Antonius Hospital
Other Study IDs: WW 22.121/NWMO22.06.013
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma; Renal Cell Carcinoma Metastatic
Keywords: decision aid; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-test: Patients with RCC receiving usual care (without use of the decision aids)
- Post-test: Patients with RCC using the decision aids
  Interventions: Other: Decision aid

INTERVENTIONS:
Other: Decision aid — Online interactive decision aid for RCC
  Groups: Post-test

SUMMARY:
The aim of this study is to evaluate the effect of two decision aids for renal cell carcinoma (RCC) on the decision-making process and the quality of the decision.

DETAILED DESCRIPTION:
Background: Treatment options for patients diagnosed with RCC depend on the stage of the disease, histopathology and patient's preferences and values regarding outcomes. For local (non-metastatic) disease, gold standard for treatment is surgical resection of the tumour. Besides this, ablative therapies or active surveillance could also be an option. For metastatic disease, targeted therapy and/or immunotherapy can be offered and new treatment options are being tested in clinical trials. The number of available treatment options for patients with RCC is increasing, but the availability of these options differs per hospital and the transparency about treatment options is limited, resulting in practice variation between hospitals.

Decision aids help patients to make decisions regarding treatment, particularly when there is not one medically superior treatment option. In this tools treatment options are explained, including outcome information such as possible side effects and benefits of therapy. Decision aids have proven to lead to increased patient knowledge, less anxiety in patients, improved health outcomes such as physical en mental health, reductions in unwarranted variation in care and costs, greater alignment of care with patients' values.

For patients with RCC, two decision aids are in development right now: one decision aid focussed on local disease and one decision aid focussed on metastatic disease. Using these decision aids, patients are encouraged to make a well-informed decision together with the healthcare professional.

Objective: To assess how the decision aids for RCC influence the quality of the decision-making processes for RCC, defined as the extent to which elements of shared decision-making (SDM) are observed.

Design, setting and participants: This study includes patients clinically diagnosed with RCC, facing a decision which is addressed in the decision aids. Study design will be a prospective multicenter pre-test post-test study.

Outcome measurements and statistical analysis: The primary endpoint of this study is the mean change in OPTION-5 score between pre-test and post-test groups. Secondary outcome measures include perceived quality of the decision-making process, quality of the decision and implementation of the decision aids.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with RCC
* Patients facing a decision which is addressed in the decision aids (T1 tumor or metastatic disease)
* Written informed consent

Exclusion Criteria:

* Patients who are not able to fill in a questionnaire or undergo an interview individually

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients clinically diagnosed with RCC
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
OPTION-5 | During consultation
  Observed patient involvement in decision-making

SECONDARY OUTCOMES:
Decisional conflict scale | Two weeks and nine weeks after consultation
  Validated scale to measure personal perceptions of uncertainty in choosing options, modifiable factors contributing to uncertainty and effective decision making.
Preparation for decision-making | Two weeks after consultation
  Validated scale that assesses the patient's perception of how useful a decision aid is in preparing the respondent to communicate with their practitioner at a consultation visit and making a health decision.
Control preference scale | Two weeks after consultation
  Validated measure of patient's preferred and actual roles in treatment decisions
SDM-Q-9 | Health care professional: directly after consultatiion, patient: two weeks after consultation
  Validated questionnaire of perceived level of shared decision-making
Knowledge check | Two weeks after consultation
  Objective assessment of patient's understanding of information relevant for the decision at stake using ten questions which can be answered as true/false/I don't know.
Implementation of the decision aids | Nine weeks after consultation
  Qualitative information about experiences with implementation and use of the decision aids will be obtained through semi-structured interviews with patients and healthcare professionals.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands